CLINICAL TRIAL: NCT04250597
Title: A Phase I Study of GNX102 in Patients With Advanced Solid Tumors
Brief Title: Study of GNX102 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Maximum tolerated dose reached; expansion phase not performed per Sponsor business decision.
Sponsor: GlycoNex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNX-001
Record Dates: First submitted 2020-01-27; First posted 2020-01-31 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor; Metastatic Cancer; Advanced Cancer; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose Escalation (Experimental): Drug: GNX102 Dose Escalation: 21 day dosing interval
  Interventions: Drug: GNX102
- Part 2 Dose Escalation (Experimental): Drug: GNX102 Dose Escalation: 7 day dosing interval
  Interventions: Drug: GNX102
- Part 3 Expansion (Experimental): Drug: GNX102 Expansion: Selected dose level(s) and schedule(s) in expanded cohort(s)
  Interventions: Drug: GNX102

INTERVENTIONS:
Drug: GNX102 — Dose Escalation
  Arms: Part 1 Dose Escalation; Part 2 Dose Escalation
Drug: GNX102 — Expansion Phase
  Arms: Part 3 Expansion

SUMMARY:
GNX102 is a humanized monoclonal antibody (mAb), an engineered biotechnology product, developed by GlycoNex that targets certain cancer cells by binding with high affinity to specific structures on cancer cells. Specifically, GNX102 binds to novel glycan structures caused by glycosylation changes in tumors.

Patients with epithelial origin cancers that have a likelihood of GNX102 targeted antigen expression based on previous studies, including colorectal, hepatocellular, non-small cell lung, gastric, breast, pancreatic, cutaneous, acral, or mucosal melanoma, esophageal, prostate, and epithelial uterine cancers, can be screened for enrollment in the study.

ELIGIBILITY:
Inclusion Criteria

The target study population consists of adult patients with advanced solid tumors that meet all of the following criteria to be enrolled into this study:

1. Age ≥ 18 years.
2. Participants with histologically confirmed solid tumors with a likelihood of expression of GNX102 targeted antigens, which are limited to:

   * colorectal
   * hepatocellular
   * non-small cell lung
   * gastric
   * breast
   * bladder
   * pancreatic
   * melanoma (cutaneous, acral, or mucosal)
   * esophageal
   * prostate
   * ovarian
   * cervical
   * epithelial uterine cancers.
3. Participant has a paraffin block of non-necrotic tumor tissue available for immunohistochemistry (IHC) analyses, to be shipped and confirmed adequate by NeoGenomics pathologist prior to initiation of treatment.
4. Advanced, unresectable (local, regionally, recurrent not amenable to curative therapy) or metastatic disease that has no standard therapeutic option with a proven clinical benefit, are intolerant to or have refused all standard of care options with demonstrated clinical benefit.
5. Expansion Phase only: Participant has measurable disease per response evaluation criteria in solid tumors (RECIST) v 1.1 criteria.
6. Eastern Cooperative Group (ECOG) performance status of 0 or 1.
7. Baseline Q-T corrected interval (QTc) interval of ≤ 480 msec using Frederica's formula.
8. Acceptable liver function:

   * Bilirubin ≤ 1.5 times upper limit of normal
   * Aspartate transaminase (serum glutamic-oxaloacetic transaminase) [AST (SGOT)] and alanine transaminase (serum glutamic-pyruvic transaminase) [ALT (SGPT)] ≤ 3 times upper limit of normal. If liver metastases are present, then ≤ 5 x upper limits of normal (ULN) is allowed, and
   * Serum albumin ≥ 2.5 g/dL.
9. Acceptable renal function, defined as calculated creatinine clearance > 30 mL/min per institution laboratory value.
10. Acceptable hematologic status:

    * Hemoglobin ≥ 8 g/dL (no packed red blood cell [PRBC] transfusions allowed within 2 weeks)
    * Absolute neutrophil count (ANC) ≥ 1500 cells/mm^3 or ≥ 1.5 x 10^9/L, and
    * Platelet count ≥ 100,000 platelets/mm^3 or ≥ 100 x 10^9/L, and
    * Absolute reticulocyte count (x10^9/L) ≤ ULN.
11. Serum haptoglobin (mg/dL) ≥ LLN.
12. Acceptable coagulation status with fibrinogen above LLN; prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time (PTT) ≤ 1.5 times upper limit of normal (may be on a stable dose of coumadin with stable INR in the therapeutic range).
13. Life expectancy of at least 3 months.
14. Signed Institutional Review Board (IRB)-approved informed consent.
15. Able and willing to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations.
16. A negative serum pregnancy test, if female of child-bearing potential.
17. For men and women of child-bearing potential, agreement to the use of at least 1 highly effective contraceptive method(s) during the study and in the 3 months following the last dose of GNX102.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from participation in this study:

1. Has any other malignancy not listed in Inclusion Criteria 2. Note: Participants with prior early-stage cervical cancer, basal cell carcinoma (BCC) or squamous cell carcinoma that has been successfully treated with curative intent and participant has been disease free for >2 years may be enrolled.
2. Has a positive polymerase chain reaction (PCR) test for active COVID-19 infection or has signs or symptoms consistent with COVID-19 in the absence of a positive PCR test within 2 weeks from date of consent.
3. Has New York Heart Association Class III or IV heart disease.
4. History of myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, within the past 6 months.
5. History of cerebral vascular accident or transient ischemic attack within the past 6 months.
6. History of primary central nervous system (CNS) tumor.
7. History of CNS metastases, unless previously treated and stable for at least 4 weeks in the absence of steroids. Participants with meningeal carcinomatosis are excluded regardless of treatment.
8. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy within 72 hours of start of therapy.
9. Active, nonmalignant gastrointestinal (GI) disease requiring treatment (such as inflammatory bowel disease, Crohn's disease, colitis) that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, which would make the participant inappropriate for entry into this study.
10. Clinical symptoms of pancreatitis within the past 28 days.
11. Known active infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C.

    * Patients with a history of hepatitis B or C are allowed if HBV deoxyribonucleic acid (DNA) or Hep C ribonucleic acid (RNA) are undetectable. Participants with hepatocellular cancer on antiviral therapy must have DNA levels ≤ 500IU/ml.
    * Participants with a history of HBV will be monitored for HBV reactivation while on study.
12. Pregnant or nursing women.
13. Treatment with radiation therapy within 14 days prior to dosing with GNX102.
14. Major surgery within 14 days prior to dosing with GNX102.
15. History of autoimmune hemolytic anemia or autoimmune thrombocytopenia.
16. Second malignancy which is considered active or requires concurrent treatment.
17. For participants with hepatocellular carcinoma

    * Ascites requiring more than 1 paracentesis per month
    * History of hepatic encephalopathy within 12 months of study entry
18. History of bleeding esophageal or gastric varices within 6 months of study entry.
19. Prior or ongoing cancer treatment, including investigational treatment within 5 half-lives or 21 days whichever is less, prior to dosing with GNX102 and 6 weeks for nitrosoureas or mitomycin C.
20. Allergies to any excipients in GNX102 (i.e., L-histidine, sucrose, Polysorbate 80).
21. Severe acute or chronic medical or psychiatric conditions or other laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, which would make the participant inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Through study completion, an average of 2 years
  If ≤ 1 of 6 patients has a dose limiting toxicity (DLT) after all previous dose testing the dose will be declared the Maximum Tolerable Dose (MTD).

SECONDARY OUTCOMES:
Antitumor activity of GNX102 | Through study completion, an average of 2 years
  To evaluate antitumor activity of GNX102 by objective radiographic assessment
AUC: Area under the concentration curve of GNX102 (μg × h/mL) | Through study completion, an average of 2 years
  To determine the AUC Area under the concentration curve of GNX102
Cmax: Maximum plasma concentration of GNX102 (μg) | Through study completion, an average of 2 years
  To determine the pharmacokinetics (PK) of GNX102
Tmax: Time to maximum plasma concentration of GNX102 (minutes) | Through study completion, an average of 2 years
  To determine the pharmacokinetics (PK) of GNX102
t1/2: Terminal phase half-life of GNX102 (minutes) | Through study completion, an average of 2 years
  To determine the pharmacokinetics (PK) of GNX102
CL: Clearance of GNX102 (L/hr) | Through study completion, an average of 2 years
  To determine the pharmacokinetics (PK) of GNX102
Vz: Apparent volume of distribution in the terminal phase of GNX102 (L) | Through study completion, an average of 2 years
  To determine the pharmacokinetics (PK) of GNX102
Number of adverse events (AEs) | Through study completion, an average of 2 years
  Dose-limiting AEs will be used to establish the MTD and the recommended dose for phase 2 studies (RP2D)
Number of toxicities | Through study completion, an average of 2 years
  Toxicities will be used to establish the MTD and the recommended dose for phase 2 studies (RP2D)

OTHER OUTCOMES:
Exploratory Outcome: GNX102 targeted antigens (counts) | Through study completion, an average of 2 years
  To explore tumor expression of GNX102 targeted antigens as a biomarker to predict toxicity or response to GNX102
Exploratory Outcome: Serum CA 19-9, CA 125, or CEA antigen levels (counts) | Through study completion, an average of 2 years
  To explore biomarkers related to participant's specific cancer type (e.g. pancreas, ovarian, or colon, respectively) to predict toxicity or response to GNX102
Exploratory Outcome: Anti-drug antibody (ADA) to GNX102 (counts) | Through study completion, an average of 2 years
  To evaluate the development of anti-drug antibody (ADA) to GNX102

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chun Yang, PhD, Study Director — President, GlycoNex, Inc.
Locations (8):
- United States (6):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Cancer Center (USC), Newport Beach, California
  - Regions Cancer Care Center, Saint Paul, Minnesota
  - Providence Cancer Institute Earle A. Chiles Research Institute, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Taiwan (2):
  - China Medical University Hospital (CMUH), Taichung
  - National Cheng Kung University Hospital (NCKUH), Tainan

IPD SHARING:
Plan to Share IPD: No